CLINICAL TRIAL: NCT03674424
Title: Avelumab as Neoadjuvant Therapy in Subjects With Urothelial Muscle Invasive Bladder Cancers
Brief Title: Avelumab as Neoadjuvant Therapy in Subjects With Urothelial Muscle Invasive Bladder Cancers (AURA Trial)
Acronym: AURA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IJB-AURA-ODN-004
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-01

CONDITIONS: Non-metastatic Muscle Invasive Bladder Cancer
MeSH Terms: interventions — avelumab; Cystectomy

STUDY DESIGN:
Intervention Model Description: Open-label, randomized study. 2 cohorts possible depending on cisplatin-eligibility. Afterwards randomization between 2 arms into the cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DD-MVAC + avelumab (Experimental): Methotrexate, vinblastine, doxorubicin and cisplatin (DD-MVAC) given in combination with Avelumab.
  DD-MVAC consists of Methotrexate 30 mg/m2 iv day 1, Vinblastine 3 mg/m2 iv day 2, Cisplatin 70 mg/m2 iv day 2 and Doxorubicin 30 mg/m2 iv day 2. Each cycle is given every 2 weeks for a maximum of 4 administrations Chemotherapy is associated with Avelumab 10 mg/kg, 1-hour intravenous (iv) infusion, given on day 2 every 2 weeks.
  Cystectomy will be performed 3 to 6 weeks after last administration of chemotherapy
  Interventions: Drug: Avelumab; Procedure: cystectomy; Combination Product: DD-MVAC
- CG+ avelumab (Experimental): Cisplatin, gemcitabine (CG) consists of Gemcitabine 1000 mg/m2 iv in day 1 and day 8 and Cisplatin 70 mg/m2 iv in day 1. Each cycle is given every 3 weeks for a maximum of 4 administrations.
  Chemotherapy is associated with Avelumab 10 mg/kg, 1-hour intravenous (iv) infusion, given on day 1 every 2 weeks Cystectomy will be performed 3 to 6 weeks after last administration of chemotherapy
  Interventions: Drug: Avelumab; Procedure: cystectomy; Combination Product: CG
- PG+ avelumab (Experimental): Paclitaxel, gemcitabine (PG) consists of Paclitaxel 80 mg/m2 iv in day 1 and day 15 and Gemcitabine 1000 mg/m2 iv in day 1 and day 15. Each cycle is repeated every 3 weeks for a maximum of 4 administrations.
  Chemotherapy is associated with Avelumab 10 mg/kg, 1-hour intravenous (iv) infusion, given on day 1 every 2 weeks Cystectomy will be performed 3 to 6 weeks after last administration of chemotherapy
  Interventions: Drug: Avelumab; Procedure: cystectomy; Combination Product: PG
- Avelumab (Experimental): Avelumab will be administered at a dose of 10 milligram per kilogram (mg/kg) 1-hour intravenous (iv) infusion once every 2 weeks. Dose reductions are not allowed.
  Avelumab will be given alone for 4 administrations. Cystectomy will be performed 2 weeks after the last administration of avelumab
  Interventions: Drug: Avelumab; Procedure: cystectomy

INTERVENTIONS:
Drug: Avelumab — Chemotherapy with or without avelumab followed by surgery
Procedure: cystectomy — Cystectomy 3 to 6 weeks after last administration of chemotherapy
Combination Product: CG — Chemotherapy 4 cycles of 3 weeks
  Arms: CG+ avelumab
Combination Product: DD-MVAC — Chemotherapy 4 cycles of 2 weeks
  Arms: DD-MVAC + avelumab
Combination Product: PG — Chemotherapy 2 cycles of 4 weeks
  Arms: PG+ avelumab

SUMMARY:
Open-label, interventional, multi-centre, randomized phase II study. Cancer studied is non-metastatic muscle invasive bladder cancer (MIBC).

Avelumab administered every 2 weeks is used as neoadjuvant therapy in subjects with urothelial muscle invasive bladder cancers in combination with standard chemotherapy or alone.

DETAILED DESCRIPTION:
Open-label, interventional, multi-centre, randomized phase II study. Cancer studied is non-metastatic muscle invasive bladder cancer (MIBC) Patients (male or female) will receive avelumab every 2 weeks in combination with standard chemotherapy or alone. There are 2 cohorts of patients.

Cohort with patients cisplatin-ineligible will receive either avelumab alone or in combination with paclitaxel-gemcitabine chemotherapy.

Cohort with patients cisplatin-eligible will receive either methotrexate, vinblastine, doxorubicine and cisplatin in combination with avelumab or cisplatin, gemcitabine in combination with avelumab.

The estimated number of subjects to screen is 183 patients for an estimated number of 166 patients enrolled for 150 evaluable patients:

26 patients in the paclitaxel, gemcitabine in combination with avelumab arm (cisplatin-ineligible patients) 26 patients in avelumab alone arm (cisplatin-ineligible patients) 49 patients in cisplatin gemcitabine + avelumab arm (cisplatin-eligible patients) 49 patients in methotrexate, vinblastine, doxorubicine and cisplatin + avelumab arm (cisplatin-eligible patients)

AVELUMAB:

Avelumab will be administered at a dose of 10 milligram per kilogram (mg/kg) 1-hour intravenous (iv) infusion once every 2 weeks. Dose reductions are not allowed.

Depending on the treatment arm, Avelumab will be given associated with chemotherapy or alone for a maximum of 4 administrations.

DD-MVAC:

DD-MVAC consists of Methotrexate 30 mg/m2 iv day 1, Vinblastine 3 mg/m2 iv day 2, Cisplatin 70 mg/m2 iv day 2 and Doxorubicin 30 mg/m2 iv day 2. Each cycle is given every 2 weeks for a maximum of 4 administrations. Pegfilgrastim 6 mg subcutaneous (SQ) 24-48 hours after completion of chemotherapy will be given.

Chemotherapy is associated with Avelumab 10 mg/kg iv given on day 2 every 2 weeks.

CG:

CG consists of Gemcitabine 1000 mg/m2 iv in day 1 and day 8 and Cisplatin 70 mg/m2 iv in day 1. Each cycle is given every 3 weeks for a maximum of 4 administrations. Pegfilgrastim 6 mg subcutaneous (SQ) 24-48 hours after completion of chemotherapy will be given.

Chemotherapy is associated with Avelumab 10 mg/kg iv given on day 1 every 2 weeks.

PG:

PG consists of Paclitaxel 80 mg/m2 iv in day 1 and day 15 and Gemcitabine 1000 mg/m2 iv in day 1 and day 15. Each cycle is repeated every 4 weeks for a maximum of 4 administrations.

Chemotherapy is associated with Avelumab 10 mg/kg i.v. given every on day 1 every 2 weeks.

For patients receiving neoadjuvant chemotherapy treatment, the surgery (cystectomy or nephroureterectomy associated to lymphadenectomy) will be performed within 3-6 weeks after the last administration of neoadjuvant chemotherapy treatment.

For patients receiving avelumab alone, the surgery will be performed 2 weeks (+7 days) after the last administration of avelumab.

Any delay in surgery (> 6 weeks after the last chemotherapy administration or >3 weeks after the last administration of avelumab alone) for any reason, needs to be discussed with the PI/Sponsor.

For all patients, neoadjuvant treatment will be stopped if there is evidence of progression of disease (by RECIST 1.1 or investigator's decision) or unacceptable toxicity according to the investigator. In this situation, the investigator will decide if it is needed to proceed directly with the surgery.

The end of study will be declared when all the following criteria will have been met:

* The study ends after last visit of the last patient remaining in the study.
* The trial is mature for the analysis of the endpoints as defined in the protocol, if the trial reaches its endpoints.
* The database has been fully cleaned and frozen for all analyses.

ELIGIBILITY:
General Inclusion Criteria:

1. Age ≥ 18 years old
2. Must have histologically confirmed muscle invasive urothelial carcinoma (transitional cell carcinoma) or urothelial carcinoma with mixed histology of the bladder, renal pelvis or ureters. Stage permitted: T2, T3 or T4a. T stage is based on the standard of care transurethral resection of the bladder tumour (TURBT) sample
3. Patients may have nodal disease (Nx, N0, N1 or N2) at imagery but there must be no evidence of distant metastases (M0)
4. Performance status 0 or 1 on the Eastern Cooperative Oncology Group (ECOG).
5. Be a medically appropriate candidate for surgery as determined by an attending urologist
6. Adequate bone marrow function as defined below:

   * Absolute neutrophil count ≥1500/µL or 1.5x109/L
   * Hemoglobin ≥ 9 g/dL
   * Platelets ≥100000/µL or 100x109/L 7)
7. Adequate liver function as defined below:

   * Serum total bilirubin ≤ 1.5 x ULN. In case of known Gilbert's syndrome < 3xUNL is allowed
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x ULN
8. Serum pregnancy test (for subjects of childbearing potential) negative within 7 days prior to study treatment administration.
9. Women of childbearing potential must agree to use one highly effective method of contraception prior study entry, during the course of the study and up to 6 months after the last administration of study treatment. Men with childbearing potential partner must agree to use condom during the course of this study and up to 6 months after the last administration of the study treatment.
10. Completion of all necessary screening procedures within 28 days prior to treatment.
11. Availability of biological material for screening and/or translational research activities
12. Signed Informed Consent form (ICF) obtained prior to any study related procedure.

    Cisplatin-eligible cohort specific criteria:
13. Glomerular filtration rate (GFR) or Creatinine Clearance≥ 60 mL/min according to the Cockcroft-Gault formula (or local institutional standard method) and
14. Peripheral neuropathy ≤ grade 1 and
15. Hearing impaired ≤ grade 1 and
16. Adequate cardiac function (Left Ventricular Ejection Fraction LVEF ≥ 55%) by MUGA (Multiple-Gated Acquisition) scan or echocardiography

    Cisplatin ineligible cohort specific criteria (if any of the following criteria):
17. Glomerular filtration rate (GFR) or Creatinine Clearance ≥ 30mL/min according to the Cockcroft-Gault formula (or local institutional standard method) or
18. Peripheral neuropathy ≥ grade 2 or
19. Hearing impaired ≥ grade 2

    Inclusion criterion specific for France:
20. Patients must be affiliated to a social security system

Exclusion Criteria:

Subjects meeting one of the following criteria are not eligible for this study:

1. Metastatic disease (M1)
2. Has had prior systemic chemotherapy, targeted small molecule therapy, or radiation therapy for urothelial carcinoma
3. Prior treatment with drug specifically targeting T-cell co-stimulation or checkpoint pathways
4. Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
5. Has an active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
6. Has had a prior organ transplantation including allogenic stem-cell transplantation.
7. Has an active infection requiring systemic therapy
8. Has a known history of Human Immunodeficiency Virus (HIV) or known acquired immunodeficiency syndrome.
9. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA is detected)
10. Has received vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines such as influenza vaccine.
11. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 28 days prior to study registration
12. History of prior invasive malignancy within 2 years (exception of adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localised prostate cancer or ductal carcinoma in situ)
13. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3)
14. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication."
15. Pregnant and/or lactating women.
16. Subject with a significant medical, neuro-psychiatric, or surgical condition, currently uncontrolled by treatment, which, in the principal investigator's opinion, may interfere with completion of the study.
17. Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade >1); however, alopecia, sensory neuropathy Grade ≤2, or other Grade ≤2 not constituting a safety risk based on investigator's judgment are acceptable.
18. Other severe acute chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behaviour; or laboratory abnormalities that may increase the risk associated with the study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

    Exclusion criterion specific for France:
19. Vulnerable persons according to the article L.1121-6 of the CSP, adults who are the subject of a measure of legal protection or unable to express their consent according to article L.1121-8 of the CSP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
To determine the pathologic complete response (ypT0/Tis ypN0) following neoadjuvant treatment in patients with non-metastatic MIBC. | during surgery
  - Outcome measure: Pathological complete response is defined as the absence of invasive carcinoma (ypT0/Tis) disease and the absence of microscopic lymph node metastases (ypN0) on the final surgical specimen.

SECONDARY OUTCOMES:
To determine the pathologic response rate (<ypT2N0) | during surgery
  Outcome measure: Pathologic response is defined as the absence of muscle invasive carcinoma (<ypT2N0 disease) on the final surgical specimen.
Assessment of the toxicity profile of regimen using the adverse events reported: NCI CTCAE v4.03 | through study completion, an average of 3 months
  Outcome measure: adverse events reported during the study according to NCI CTCAE v4.03
Assessment of local or distant recurrence | at 12 and 36 months after surgery (or at 12 and 36 months after last treatment dose if no surgery was performed)
  Outcome measure: invasive disease-free survival (iDFS) rate. iDFS period is defined as a time between the surgery (or last treatment dose if no surgery) and the date of diagnosis of local or distant recurrence, or secondary primary malignancy
Assessment of overall survival | minimum 36 months FU after surgery (or after last treatment dose if no surgery).
  overall survival (OS) rate. Overall survival is defined as a time between the surgery (or last treatment dose if no surgery) and the day of death (due to any causes) or day of last news

CONTACTS AND LOCATIONS:
Locations (10):
- Belgium (6):
  - UZAntwerpen, Edegem, Antwerpen
  - Centre Hospitalier Universitaire et Psychiatrique de Mons-Borinage, Mons, Hainaut
  - Institut Jules Bordet, Brussels
  - Grand Hôpital de Charleroi, Gilly
  - CHU de Liège Sart Tilman, Liège
  - CHU Namur - Sainte Elisabeth, Namur
- France (4):
  - Centre Oscar Lambret, Lille
  - Groupe Hospitalier Paris Saint Joseph, Paris
  - Hôpital Saint Louis, Paris
  - Hôpitaux universitaires de Strasbourg, Strasbourg

REFERENCES:
- [Derived] Blanc J, Carnot A, Barthelemy P, Casert V, Sautois B, Van den Brande J, Vanhaudenarde V, Staudacher L, Seront E, Debien V, Ameye L, Kotecki N, Rothe F, Rorive S, Fantoni JC, Tricard T, Roumeguere T, Awada A, Martinez Chanza N. Avelumab-based neoadjuvant therapy in patients with muscle-invasive bladder cancer (AURA Oncodistinct-004): a phase 2 multicenter clinical trial. J Immunother Cancer. 2025 May 24;13(5):e012045. doi: 10.1136/jitc-2025-012045. PMID 40413024
- [Derived] Martinez Chanza N, Soukane L, Barthelemy P, Carnot A, Gil T, Casert V, Vanhaudenarde V, Sautois B, Staudacher L, Van den Brande J, Culine S, Seront E, Gizzi M, Albisinni S, Tricard T, Fantoni JC, Paesmans M, Caparica R, Roumeguere T, Awada A. Avelumab as neoadjuvant therapy in patients with urothelial non-metastatic muscle invasive bladder cancer: a multicenter, randomized, non-comparative, phase II study (Oncodistinct 004 - AURA trial). BMC Cancer. 2021 Dec 2;21(1):1292. doi: 10.1186/s12885-021-08990-3. PMID 34856936